CLINICAL TRIAL: NCT06671288
Title: "Effects of Balloon-blowing Exercises With Abdominal & Lumbar Core Muscle Activation Position Among Smokers"
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/27
Record Dates: First submitted 2024-09-20; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-08

CONDITIONS: Smoking
Keywords: dysnea; Cigarette smoking; spirometry; Quality of life
MeSH Terms: conditions — Smoking; Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups. One group will receive (interventional group) balloon-blowing exercises with abdominal & lumbar core muscles activation position.
  and the other group (control group) will receive Diaphragmatic breathing exercise.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Patients in this group will receive balloon -blowing exercise with abdominal & lumbar core muscle activation position Total 4 weeks protocol. Three sessions per week will be supervised by physical therapist.
  Interventions: Other: Balloon-blowing exercises with abdominal & lumbar core muscle activation position.
- Control group (Active Comparator): Patients will receive diaphragmatic breathing exercises. Total 4 weeks protocol.
  Before and after 4 weeks pre and post interventional values will be taken.
  Interventions: Other: Diaphragmatic breathing exercise

INTERVENTIONS:
Other: Balloon-blowing exercises with abdominal & lumbar core muscle activation position. — Patients in this group will recieve Balloon-blowing exercises with abdominal and lumbar core muscles activation position Total 4 weeks protocol will be followed in which 3 sessions per week will be supervised by physical therapist.
  FREQUENCY: 3 times a week, INTENSITY : Moderate, TIME: 4 sets of balloon-blowing with 1 min rest (30 mins) TYPE: Balloon-blowing with abdominal & lumbar core muscle activation position, DURATION : 4 weeks
  Arms: Interventional group
Other: Diaphragmatic breathing exercise — Participants in this group will only be receiving diaphragmatic breathing exercise for 4 weeks. FREQUENCY: 3 times a week , INTENSITY: Moderate, TIME: 4 sets of diaphragmatic breathing with 1 min rest, TYPE: Diaphragmatic breathing, DURATION: 4 weeks
  Arms: Control group

SUMMARY:
The principle function of the lungs is the facilitation of the gaseous exchange, commonly referred as respiratory or breathing. Cigarette smoking has detrimental effects on nearly every organ in the body, leading to a higher incidence of diseases and contributing to a gradual deterioration of the smoker's health.Cigarette smoking has detrimental effects on nearly every organ in the body, leading to a higher incidence of diseases and contributing to a gradual deterioration of the smoker's health.

Cigarette smoking is linked to mild airway obstruction and a deceleration in the growth of lung function.Performing balloon-blowing exercises with abdominal and lumbar core muscles activation position leads to an improvement on pulmonary function and quality of life in smokers.

DETAILED DESCRIPTION:
Cigarette smoking has detrimental effects on nearly every organ in the body, leading to a higher incidence of diseases and contributing to a gradual deterioration of the smoker's health, including a progressive impairment of lung function. Cigarette smoking is linked to mild airway obstruction and a deceleration in the growth of lung function.

Smokers may experience inflammation and narrowing of their airways, resulting in increased resistance to the outward flow of air during exhalation. This restriction in airflow can negatively impact respiratory parameters, exercise tolerance, and overall quality of life.

Performing balloon-blowing exercises with abdominal and lumbar core muscles activation position leads to an improvement on pulmonary function and quality of life in smokers.

ELIGIBILITY:
Inclusion Criteria:

* Adults: aged (25-59 years)
* Gender: Both males and females
* Grade1- Grade 4 on Modified MRC dyspnea scale
* COPD classes (mild, moderate ) according to GOLD COPD Guidelines
* Participating voluntarily and follow the instructions & performing
* The number of packs of cigarettes smoked per day by the number of years the person has smoked.

  1. pack yr = 20 cig/day x 1 yrs
  2. pack yr = 20 cig/day x 2 yrs

Exclusion criteria:

* Severe cases of obstruction like Severe asthma & status asthmaticus, Severe COPD, bullous emphysema for pneumothorax.
* Any congenital deformities of chest wall, Demonstrated neuromuscular or neurological deficit/disease of chest wall
* Other serious Cardiopulmonary diseases including pulmonary embolism, pulmonary ----Hypertension, Active TB, pneumonias or other acute illnesses
* Any recent cardiothoracic or abdominal surgery, trauma or injury
* Pregnancy
* Any psychiatric illnesses

Ages: 25 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
FVC (forced vital capacity): | 4 weeks
  FVC (forced vital capacity): The amount of air that can be maximum forcefully be exhaled after taking deep breath.
FEV1 | 4 weeks
  FEV1(Forced expiratory volume in 1 second): The volume of air that is forcefully exhaled in one second.
FEV1/FVC | 4 weeks
  FEV1/FVC: The ratio of the forced expiratory volume in the first one second to the forced vital capacity of the lungs.
PEF (Peak expiratory flow) | 4 Weeks
  PEF( Peak expiratory flow): Measurement of the highest speed at which a individual can exhale air from their lungs after a full inhalation.
Dyspnea | 4 Weeks
  Evaluation will be done using mMRC dyspnea scale (0-4). 0 I only get breathless with strenuous exercise
  1. I get short of breath when hurrying on level ground or walking up a slight hill
  2. On level ground, I walk slower than people of the same age because of breathlessness, or have to stop for breath when walking at my own pace
  3. I stop for breath after walking about 100 yards [91 meters] or after a few minutes on level ground
  4. I am too breathless to leave the house or I am breathless when dressing
Quality of life of participant | 4 weeks
  Quality of life questionnaire (SF-36) will be used to evaluate smokers QOLSF-36 Questionnaire (0-100). Each question carries equal weight the lower the score the more the disability. The higher the score the lesser the disability.
  0: Maximum disability 100: No disability
Oxygen saturation | 4 weeks
  Pulse oximeter will be used to measure oxygen saturation

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan